CLINICAL TRIAL: NCT01481116
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-875 25 mg and 50 mg Compared to Glimepiride When Used in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of TAK-875 Compared to Glimepiride When Used With Metformin in Participants With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_304; 2011-001731-24 (EudraCT Number); U1111-1124-2296 (Registry Identifier: WHO); TAK-875_304CTIL (Other: Israel MOH); DOH-27-0512-3913 (Registry Identifier: SANCTR); 11-057 (Registry Identifier: ROCTR); NMRR-11-882-10318 (Registry Identifier: NMRR); HKCTR-1616 (Registry Identifier: HKUCTR); 262 (Registry Identifier: RoPCCT); 12/WA/0245 (Registry Identifier: NRES)
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAK-875 25 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 50 mg QD (Experimental)
  Interventions: Drug: TAK-875
- Glimepiride 1-2 mg QD (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: TAK-875 — TAK-875 25 mg, tablets, orally, once daily and metformin ≥1500 mg or Maximum Tolerated Dose (MTD) for up to 104 weeks.
  Arms: TAK-875 25 mg QD
Drug: TAK-875 — TAK-875 50 mg, tablets, orally, once daily and metformin ≥1500 mg or MTD for up to 104 weeks.
  Arms: TAK-875 50 mg QD
Drug: Glimepiride — Glimepiride 1 mg, tablets, orally, once daily (up-titrated to 2 mg after 1 week of treatment. Up-titrated to a maximum of 6 mg in 2 mg increments/down titrated if recurrent (or severe) hypoglycemia occurs) and metformin ≥1500 mg or MTD for up to 104 weeks.
  Arms: Glimepiride 1-2 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-875, once daily (QD), plus metformin compared to glimepiride plus metformin in participants with type 2 diabetes mellitus (T2DM).

The purpose of this study is to determine the efficacy and safety of TAK-875, once daily (QD), plus metformin compared to glimepiride plus metformin in participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) has increased dramatically throughout the world over the past decades despite the availability of several different treatment options. Current pharmacologic treatments include insulin, thiazolidinediones, sulfonylureas, metformin, dipeptidyl-peptidase-4 (DPP-4) inhibitors, and glucagon-like peptide-1 (GLP-1) mimetics. A number of these treatments are associated with clinically important side effects such as low blood sugar (hypoglycemia), weight gainflud retention, exaggeration of pre-existent heart failure, and gastrointestinal side effects. These side effects and the disadvantages associated with many of the currently available antidiabetic agents can reduce compliance and limit their long-term use.

Insulin is a hormone that is produced by the body to regulate blood sugar (glucose). In individuals with T2DM, the insulin produced by the body does not effectively control the amount of sugar in the bloodstream. If not properly managed, T2DM may cause elevated blood sugar levels (hyperglycemia) and ultimately result in serious health problems.

In response to this problem, Takeda is developing TAK-875 (an investigational drug) as an addition to diet and exercise to improve blood sugar control in patients with T2DM. TAK-875 may affect the production of insulin and may improve how the body uses the sugar in the blood.

The aim of this study is to find out if TAK-875, when taken for approximately 2 years in combination with current diabetes medicine (called metformin), is safe and effective at helping people with T2DM control their high blood sugar when compared to glimepiride (a type of medication called a sulfonylurea). The study is being done to find out if the combination of TAK-875 plus metformin works as well as the combination of glimepiride plus metformin.

Approximately 2430 patients worldwide aged 18 or over with T2DM, will take part in this study and will be involved in the study for up to 110 or 120 weeks.

TAK-875 is being developed at Takeda Global Research and Development, Inc. as an adjunct to diet and exercise to improve glycemic control in participants with T2DM.

This study will investigate TAK-875 in participants with type 2 diabetes mellitus whose blood sugar level is inadequately controlled with metformin monotherapy.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is male or female and 18 years of age or older with a historical diagnosis of T2DM.
4. The participant meets one of the following criteria:

   1. The participant has an HbA1c level ≥7.0 and <10.0%, and has been on a stable daily dose of ≥1500 mg (or documented MTD) of metformin for at least 2 months prior to Screening. This participant will immediately enter the Placebo Run-in Period, or;
   2. The participant has an HbA1c level ≥ 7.5 and <10.5%, and has been on a stable daily dose of <1500 mg of metformin without documented MTD for at least 2 months prior to Screening. After completing the Screening Visit, this participant will have their metformin dose immediately increased to ≥1500 mg (or MTD) for an 8-week Titration Period. Following this 8-week period, the participant must qualify for entry into the Placebo Run-in Period by completing the Week -3 procedures and having an HbA1c concentration ≥7.0 and <10.0%.
5. The participant has had no treatment with antidiabetic agents other than metformin within 2 months prior to Screening (Exception: if a participant has received other antidiabetic therapy for ≤7 days within the 2 months prior to Screening).
6. The participant has a body mass index (BMI) of ≤45 kg/m2 at Screening.
7. Participants regularly using other, non-excluded medications, must be on a stable dose for at least 4 weeks prior to Screening. However, PRN (as needed) use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
8. The participant is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete participant diaries.

Additional Inclusion Criteria Prior to Randomization

1. The participant has an HbA1c concentration ≥7.0% and <10.0%, and a FPG ≤270 mg/dL (15.0 mmol/L) at the Week -1 Visit. (If the subject does not qualify for randomization based on these criteria, the assessment may be repeated weekly, for a maximum of 2 additional weeks).
2. The participant's compliance with the single-blind study medication during the Placebo Run-in Period is at least 75% and does not exceed 125% based on tablet/capsule counts performed by the study staff.
3. A female participant of childbearing potential must have a negative urine hCG pregnancy test at Baseline (Day 1) prior to Randomization and prior to administration of the first dose of double-blind study medication.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to Screening or has received an investigational antidiabetic drug within the 3 months prior to Screening.
2. The participant has been randomized into a previous TAK-875 study
3. The participant is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
4. The participant donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. The participant has a hemoglobin ≤12 g/dL (≤120 gm/L) for males and ≤10 g/dL (≤100 gm/L) for females at Screening.
6. The participant has a systolic blood pressure ≥160 mm Hg or diastolic pressure ≥95 mm Hg at Screening (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement).
7. The participant has history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
8. The participant has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0x upper limit of normal (ULN) at Screening.
9. The participant has a total bilirubin level greater than the ULN at Screening. Exception: if a participant has documented Gilbert's Syndrome the participant will be allowed with an elevated bilirubin level per the investigator's discretion.
10. The participant has a serum creatinine ≥1.5 mg/dL(males) and ≥1.4 mg/dL(females) and/or estimated glomerular filtration rate (GFR) <60 mL/min/1.73m2 at Screening.
11. The participant has uncontrolled thyroid disease.
12. The participant has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. The participant has had gastric banding, or gastric bypass surgery within one year prior to Screening.
14. The participant has a known history of infection with human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
15. The participant had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior to or at Screening.
16. The participant has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to any component of TAK-875, metformin, or glimepiride.
17. The participant has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
18. The participant received excluded medications prior to Screening or is expected to receive excluded medication.
19. If female, the participant is pregnant (confirmed by laboratory testing, i.e., serum/urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
20. The participant is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
21. The participant has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Additional Exclusion Criteria Prior to Randomization

1. The participant has received excluded medications listed in the protocol during the Placebo Run-in Period (topical and inhaled corticosteroids are allowed).
2. The participant has a systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥95 mm Hg at Baseline (Day 1) (If the subject meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement and decision will be made based on the second measurement).
3. The participant has a serum creatinine ≥1.5 mg/dL(≥133µmol/L) [males] and ≥1.4 mg/dL (≥124 µmol/L) [females] and/or estimated glomerular filtration rate (GFR) <60 mL/min/1.73m2 at Visit 3 (Schedule B subjects only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2454 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Takeda
Locations (226):
- United States (46):
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Goodyear, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Long Beach, California
  - Mission Hills, California
  - North Hollywood, California
  - Norwalk, California
  - Pismo Beach, California
  - Bradenton, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Hialeah, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Decatur, Georgia
  - Avon, Indiana
  - Topeka, Kansas
  - Oxon Hill, Maryland
  - Flint, Michigan
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Elizabeth, New Jersey
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Maumee, Ohio
  - Oklahoma City, Oklahoma
  - Greer, South Carolina
  - Spartanburg, South Carolina
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Hampton, Virginia
  - Manassas, Virginia
- Argentina (6):
  - Buenos Aires, Ciudad Autonoma Buenos Aires
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Corrientes, Corrientes Province
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - Córdoba
- Australia (5):
  - Canberra, Australian Capital Territory
  - Brookvale, New South Wales
  - Mosman, New South Wales
  - Woy Woy, New South Wales
  - Canberra
- Bulgaria (8):
  - Blagoevgrad
  - Gabrovo
  - Pleven
  - Plovdiv
  - Sevlievo
  - Sofia
  - Stara Zagora
  - Varna
- Canada (10):
  - Victoria, British Columbia
  - Oakville, Ontario
  - Ottawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Longueuil, Quebec
  - Mirabel, Quebec
  - Pointe-Claire, Quebec
  - Saint-Laurent, Quebec
- Colombia (2):
  - Bogotá
  - Medellín
- Czechia (13):
  - Benátky nad Jizerou
  - Brno
  - Choceň
  - České Budějovice
  - Jindřichův Hradec
  - Mariánské Lázně
  - Olomouc
  - Ostrava
  - Ostrava - Moravska Ostrava
  - Ostrava - Vitkovice
  - Prague
  - Praha 4 - Krc
  - Znojmo
- Estonia (6):
  - Paide
  - Rakvere
  - Saku
  - Tallinn
  - Tartu
  - Võru
- Hong Kong (2):
  - Hong Kong
  - New Territories
- Israel (17):
  - Ashkelon
  - Beer Yaakov
  - Beersheba
  - Giv‘atayim
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Raanana
  - Ramat Gan
  - Rehovot
  - Rishon LeZiyyon
  - Safed
  - Tel Aviv
- Latvia (6):
  - Jelgava
  - Limbaži
  - Ogre
  - Riga
  - Talsi
  - Valmiera
- Lithuania (4):
  - Alytus
  - Kaunas
  - Klaipėda
  - Vilnius
- Malaysia (9):
  - Kuala Lumpur, Kuala Lumpur
  - Malacca, Melaka
  - Ipoh, Perak
  - Taiping, Perak
  - Taiping, Perak, Perak
  - Putrajaya, Putrajaya
  - Petaling Jaya, Selangor
  - Terengganu, Terengganu
  - Terengganu
- Mexico (2):
  - Mexico City, Mexico City
  - Cuernavaca, Morelos
- New Zealand (7):
  - Auckland
  - Christchurch
  - Hamilton
  - Palmerston North
  - Rotorua
  - Tauranga
  - Wellington
- Philippines (7):
  - Cebu City
  - Davao City
  - Iloilo City
  - Lipa City
  - Quezon City
  - Tarlac City
  - Taytay
- Poland (20):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Grodzisk Mazowiecki
  - Kamieniec Ząbkowicki
  - Katowice
  - Lodz
  - Lublin
  - Oświęcim
  - Parczew
  - Poznan
  - Puławy
  - Płock
  - Ruda Śląska
  - Rzeszów
  - Sopot
  - Torun
  - Wroclaw
  - Zgierz
  - Łęczyca
- Romania (9):
  - Bacau
  - Baia Mare
  - Bucharest
  - Constanța
  - Iași
  - Oradea
  - Ploieşti
  - Târgu Mureş
  - Timișoara
- Russia (7):
  - Kazan'
  - Kemerovo
  - Krasnoyarsk
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Yaroslavl
- South Africa (12):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Krugersdorp, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Middelburg, Mpumalanga
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Stellenbosch, Western Cape
  - Worcester, Western Cape
- Taiwan (5):
  - Chia-Yi City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei
- Ukraine (12):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Luhansk
  - Lviv
  - Mykolayiv
  - Poltava
  - Ternopil
  - Vinnytsia
  - Zaporizhzhia
- United Kingdom (11):
  - Cardiff, Cardiff
  - Cheadle, Cheshire
  - Plymouth, Devon
  - Hull, East Riding of Yorkshire
  - Bexhill-on-Sea, East Sussex
  - Watford, Hertfordshire
  - Thornton-Cleveleys, Lancashire
  - Liverpool, Merseyside
  - Northwood, Middlesex
  - Bath, Somerset
  - Swansea, South Glamorgan

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 291 sites in Argentina, Australia, Bulgaria, Canada, Colombia, Czech Republic, Estonia, Hong Kong, Israel, Latvia, Lithuania, Malaysia, Mexico, New Zealand, Philippines, Poland, Romania, the Russian Federation, South Africa, Taiwan, Ukraine, the United Kingdom and the United States from 06 November 2011 to 24 April 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who were inadequately controlled while receiving metformin alone were enrolled in 1 of 3 treatment groups as follows: glimepiride; TAK-875 25 milligram (mg); TAK-875 50 mg.
Groups:
- Glimepiride: TAK-875 placebo-matching tablets, orally, once daily and glimepiride 1 mg, over-encapsulated capsules, orally, once daily for 1 week followed by up-titration in 2 mg increments up to 6 mg, orally, once daily along with metformin greater than or equal to (>=)1500 mg per day or maximum tolerated dose, tablets, orally for up to 104 weeks. Glimepiride dose could be down-titrated from 6 mg in case of recurrent or severe hypoglycemia.
- TAK-875 25 mg: TAK-875 25 mg, tablets, orally, once daily and glimepiride placebo-matching capsules, orally, once daily along with metformin >=1500 mg per day or maximum tolerated dose, tablets, orally for up to 104 weeks.
- TAK-875 50 mg: TAK-875 50 mg, tablets, orally, once daily and glimepiride placebo-matching capsules, orally, once daily along with metformin >=1500 mg per day or maximum tolerated dose, tablets, orally for up to 104 weeks.
Period: Overall Study
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Started | 824 | 817 | 813
Treated | 822 | 816 | 813
Completed | 0 | 0 | 0
Not Completed | 824 | 817 | 813
Not completed — Adverse Event | 26 | 26 | 42
Not completed — Major Protocol Deviation | 3 | 7 | 1
Not completed — Lost to Follow-up | 8 | 12 | 11
Not completed — Withdrawal by Subject | 37 | 33 | 37
Not completed — Study Termination | 730 | 729 | 713
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Lack of Efficacy | 3 | 3 | 1
Not completed — Contraindications | 1 | 1 | 0
Not completed — Other | 1 | 1 | 0
Not completed — Participant Started Taking Glipizide | 1 | 0 | 0
Not completed — Participant Moved Out of Area | 2 | 0 | 1
Not completed — Participant Moved Out of Country | 1 | 0 | 1
Not completed — Investigator Decision | 3 | 2 | 1
Not completed — Sponsor Decision | 0 | 1 | 3
Not completed — Non-Compliant With Study Drug | 0 | 1 | 1
Not completed — Investigator's Discretion | 2 | 0 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Hypoglycemic Event | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg | Total
Number analyzed (Participants) | 824 | 817 | 813 | 2454
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.56) | 56.8 (9.34) | 56.6 (9.81) | 56.9 (9.57)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 637 | 646 | 648 | 1931
  >=65 years | 187 | 171 | 165 | 523
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 428 | 422 | 362 | 1212
  Male | 396 | 395 | 451 | 1242
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 68 | 66 | 70 | 204
  Non-Hispanic or Latino | 105 | 110 | 106 | 321
  Not Available | 651 | 641 | 637 | 1929
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 8 | 20 | 12 | 40
  Asian | 101 | 99 | 93 | 293
  Black or African American | 62 | 70 | 77 | 209
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7 | 14
  White | 617 | 598 | 601 | 1816
  Multiracial | 33 | 26 | 23 | 82
Region of Enrollment [Number; unit: participants]
  Argentina | 37 | 39 | 37 | 113
  Australia | 4 | 2 | 3 | 9
  Bulgaria | 17 | 18 | 16 | 51
  Canada | 42 | 40 | 39 | 121
  Colombia | 2 | 0 | 1 | 3
  Czech Republic | 31 | 31 | 31 | 93
  Estonia | 12 | 12 | 12 | 36
  Hong Kong | 9 | 10 | 10 | 29
  Israel | 50 | 50 | 50 | 150
  Latvia | 15 | 14 | 14 | 43
  Lithuania | 21 | 23 | 22 | 66
  Malaysia | 17 | 16 | 17 | 50
  Mexico | 14 | 14 | 15 | 43
  New Zealand | 15 | 14 | 15 | 44
  Philippines | 39 | 38 | 37 | 114
  Poland | 64 | 66 | 63 | 193
  Romania | 52 | 52 | 51 | 155
  Russian Federation | 26 | 26 | 26 | 78
  South Africa | 83 | 81 | 83 | 247
  Taiwan, Province Of China | 11 | 11 | 12 | 34
  Ukraine | 80 | 80 | 79 | 239
  United Kingdom | 18 | 16 | 17 | 51
  United States | 165 | 164 | 163 | 492
Height [Mean (Standard Deviation); unit: centimeter (cm)] — For this outcome measure, number of participants evaluable were 823, 817 and 813 for each arm, respectively.
  centimeter (cm) | 166.2 (10.66) | 166.2 (10.23) | 167.3 (10.19) | 166.6 (10.37)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — For this outcome measure, number of participants evaluable were 822, 816 and 813 for each arm, respectively.
  kilogram (kg) | 86.95 (18.415) | 87.35 (18.283) | 88.37 (18.796) | 87.55 (18.501)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — For this outcome measure, number of participants evaluable were 821, 816 and 813 for each arm, respectively.
  kilogram per square meter (kg/m^2) | 31.34 (5.334) | 31.50 (5.253) | 31.43 (5.403) | 31.42 (5.329)
Smoking Classification [Number; unit: participants]
  Never smoked | 552 | 533 | 502 | 1587
  Current smoker | 114 | 143 | 126 | 383
  Ex-smoker | 158 | 141 | 185 | 484
Baseline Glycosylated Hemoglobin (HbA1c) Category [Number; unit: participants]
  < 8.5 percent (%) | 584 | 584 | 592 | 1760
  >=8.5% | 238 | 232 | 221 | 691
  Not Available | 2 | 1 | 0 | 3
Duration of Diabetes [Mean (Standard Deviation); unit: years] — For this outcome measure, number of participants evaluable were 823, 817 and 812 for each arm, respectively.
  years | 6.372 (5.293) | 6.566 (5.132) | 5.995 (4.711) | 6.312 (5.056)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Weeks 78 and 104
Description: The change in the value of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) to be collected at Weeks 78 and 104 relative to baseline.
Time Frame: Baseline and Weeks 78 and 104
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline and at least 1 post- baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 62 | 61 | 66
percentage of glycosylated hemoglobin
  Baseline | 8.00 (0.814) | 8.01 (0.777) | 7.99 (0.792)
  Change at Week 78 | -0.80 (0.957) | -0.82 (0.865) | -0.98 (0.834)
  Change at Week 104 | NA (NA) — Data was not reported as none of the participants had data for this arm at this time point. | -1.03 (1.159) | 0.03 (0.603)

2. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: Participants were provided diaries to document any hypoglycemic events that occurred between study visits. Any experience of hypoglycemic signs and symptoms (regardless of the blood glucose value by glucometer) or had a blood glucose value less than or equal to (<=) 70 milligram per deciliter (mg/dL) (3.9 millimole per liter (mmol/L) by glucometer (regardless of symptoms) were to be recorded.
Time Frame: Day 1 up to Weeks 78 and 104
Population: Safety analysis set included all participants who received at least 1 dose of double-blind study medication. Participants were analyzed according to the study medication they received.
Measure: Number; unit: percentage of participants
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 822 | 816 | 813
percentage of participants
  Day 1 up to Week 78 | 30.2 | 5.4 | 5.3
  Day 1 up to Week 104 | 30.2 | 5.4 | 5.3
Statistical Analysis 1: Comparison: Glimepiride vs TAK-875 25 mg; Day 1 up to Week 78: Odds Ratios, corresponding confidence interval, and p-values were calculated using logistic regression with factors for treatment, country, schedule and baseline HbA1c value; Test type: Superiority or Other; p < 0.001, Regression, Logistic — The testing procedure at 2-sided significance level of 0.025 was as follows: 1) TAK-875 25 mg vs. glimepiride, 2) TAK-875 50 mg plus metformin vs. glimepiride. If P-value was not greater than 0.025 at Step 1, then Step 2 was carried out; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.09 to 0.18]
Statistical Analysis 2: Comparison: Glimepiride vs TAK-875 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.09 to 0.18]
Statistical Analysis 3: Comparison: Glimepiride vs TAK-875 25 mg; Day 1 up to Week 104: Odds Ratios, corresponding confidence interval, and p-values were calculated using logistic regression with factors for treatment, country, schedule and baseline HbA1c value; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.09 to 0.18]
Statistical Analysis 4: Comparison: Glimepiride vs TAK-875 50 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.09 to 0.18]

3. Secondary Outcome: Change From Baseline in Body Weight at Weeks 78 and 104
Description: The change between the body weight to be collected at Weeks 78 and 104 relative to baseline.
Time Frame: Baseline and Weeks 78 and 104
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline and at least 1 post- baseline value during the double-blind treatment period. Data for body weight was not available at Week 104 due to early termination of the study.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 51 | 44 | 55
kg
  Baseline | 84.32 (0.981) | 84.55 (1.003) | 85.67 (0.995)
  Change at Week 78 | 1.24 (0.492) | -0.07 (0.524) | -0.21 (0.487)
Statistical Analysis 1: Comparison: Glimepiride vs TAK-875 25 mg; Change at Week 78; Test type: Superiority or Other; p = 0.065, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; Treatment, schedule and visit-by-treatment interaction as fixed factors and with baseline value and baseline value by visit interaction as covariates; Least Squares Mean Difference = -1.31, 95% CI 2-sided [-2.70 to 0.08], Standard Error of Mean 0.707
Statistical Analysis 2: Comparison: Glimepiride vs TAK-875 50 mg; Change at Week 78; Test type: Superiority or Other; p = 0.034, Mixed Model Repeated Measures — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = -1.44, 95% CI 2-sided [-2.78 to -0.11], Standard Error of Mean 0.678

4. Secondary Outcome: Change From Baseline in HbA1c at Weeks 26 and 52
Description: The change in the value of HbA1c collected at Weeks 26 and 52 relative to baseline.
Time Frame: Baseline and Weeks 26 and 52
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline and at least 1 post- baseline value during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 652 | 645 | 641
percentage of glycosylated hemoglobin
  Week 26 | -0.91 (0.039) | -0.63 (0.039) | -0.81 (0.039)
  Week 52 | -0.78 (0.043) | -0.65 (0.044) | -0.81 (0.043)

5. Secondary Outcome: Percentage of Participants With HbA1c <7%
Time Frame: Weeks 26, 52, 78 and 104
Population: FAS included all randomized subjects who received at least 1 dose of double-blind study medication and who had a baseline and at least 1 post- baseline value during the double-blind treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 652 | 645 | 641
percentage of participants
  Week 26 | 51.8 | 38.3 | 48.7
  Week 52 | 47.8 | 43.3 | 54.5
  Week 78 | 45.2 | 37.7 | 54.5
  Week 104 | NA — Data was not reported as none of the participants had data for this arm at this time point. | 33.3 | 33.3

6. Secondary Outcome: Percentage of Participants With HbA1c <7% for Participants Who Did Not Report Hypoglycemia
Time Frame: Weeks 26, 52, 78 and 104
Population: Data for this outcome measure was not analyzed as prespecified in the protocol.
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Weeks 26, 52, 78 and 104
Description: The change between the fasting plasma glucose value to be collected at Weeks 26, 52, 78 and 104 relative to baseline.
Time Frame: Baseline and Weeks 26, 52, 78 and 104
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Number analyzed (Participants) | 652 | 816 | 813
milligram per deciliter (mg/dL)
  Baseline | 164.5 (41.25) | 165.2 (38.45) | 163.7 (38.65)
  Change at Week 26 | -19.5 (41.90) | -17.4 (34.67) | -23.0 (31.99)
  Change at Week 52 | -19.8 (40.81) | -19.3 (36.85) | -23.7 (33.78)
  Change at Week 78 | 0.0 (41.87) | -17.6 (30.03) | -21.4 (41.27)
  Change at Week 104 | NA (NA) — Data was not reported as none of the participants had data for this arm at this time point. | -24.0 (1.41) | -32.0 (17.58)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events started after first dose of study drug and no more than 30 days for a serious adverse event after the last dose of study drug. Time of individual participant follow-up ranged from 1 to 735 days.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Glimepiride | TAK-875 25 mg | TAK-875 50 mg
Serious Adverse Events (participants affected / at risk) | 63/822 | 41/816 | 58/813
Other Adverse Events (participants affected / at risk) | 334/822 | 337/816 | 323/813
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glimepiride (N=822) | TAK-875 25 mg (N=816) | TAK-875 50 mg (N=813)
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 4
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Retinal artery thrombosis (Eye disorders) | 0 | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 3 | 2 | 3
Chest discomfort (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 4
Appendicitis (Infections and infestations) | 0 | 0 | 2
Peritonitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0
Keratitis fungal (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Linitis plastica (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glimepiride (N=822) | TAK-875 25 mg (N=816) | TAK-875 50 mg (N=813)
Diarrhoea (Gastrointestinal disorders) | 28 | 35 | 36
Blood creatine phosphokinase increased (Investigations) | 26 | 15 | 17
Dizziness (Nervous system disorders) | 20 | 16 | 9
Nausea (Gastrointestinal disorders) | 18 | 18 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 13 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 26 | 16
Urinary tract infection (Infections and infestations) | 28 | 22 | 29
Bronchitis (Infections and infestations) | 25 | 22 | 25
Headache (Nervous system disorders) | 47 | 42 | 34
Pharyngitis (Infections and infestations) | 16 | 10 | 17
Nasopharyngitis (Infections and infestations) | 44 | 38 | 45
Upper respiratory tract infection (Infections and infestations) | 55 | 73 | 59
Influenza (Infections and infestations) | 38 | 31 | 31
Hypertension (Vascular disorders) | 47 | 28 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 28 | 22
Alanine aminotransferase increased (Investigations) | 17 | 22 | 24
Hyperuricaemia (Metabolism and nutrition disorders) | 19 | 12 | 15
Fatigue (General disorders) | 10 | 6 | 17
Dyslipidaemia (Metabolism and nutrition disorders) | 15 | 10 | 17
Gastroenteritis (Infections and infestations) | 11 | 12 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 33 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.